CLINICAL TRIAL: NCT05559892
Title: Conditional Cash Transfer Intervention to Improve Health Outcomes Among Inner-City African Americans With T2DM
Brief Title: Conditional Cash Transfer Intervention to Improve T2DM
Acronym: DMCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jennifer Annette Campbell, Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1K01DK131319 (NIH)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes-Tailored CCTs (DM-CCT) Intervention (Experimental): Participants randomized to DM-CCT will receive cash transfers of $500 per month for 6 months, but the cash transfers will be conditional on attending a 60-minute diabetes education/skills training (30 minutes) and stress/coping (30 minutes) session delivered by trained nurses every 2 weeks for 6 months (12 sessions). Therefore, they will only receive cash transfer payments if they attend two sessions per month.
  Interventions: Behavioral: DM-CCT
- Unconditional Cash Transfer-UCTs Intervention (Active Comparator): Participants randomized to UCT will receive cash transfers of $500 per month for 6 months, but there will be no conditions attached. Therefore, they will receive cash transfer payments every month. However, to control for content and attention, participants will receive mailed version of the diabetes education/skills training materials every two weeks on the same schedule as the DM-CCT telephone sessions.
  Interventions: Behavioral: DM-UCT

INTERVENTIONS:
Behavioral: DM-CCT — Participants randomized to DM-CCT will receive cash transfers of $500 per month for 6 months, but the cash transfers will be conditional on attending a 60-minute diabetes education/skills training (30 minutes) and stress/coping (30 minutes) session delivered by trained nurses every 2 weeks for 6 months (12 sessions).
  Arms: Diabetes-Tailored CCTs (DM-CCT) Intervention
Behavioral: DM-UCT — Participants randomized to UCT will receive cash transfers of $500 per month for 6 months, but there will be no conditions attached. Therefore, they will receive cash transfer payments every month. However, to control for content and attention, participants will receive mailed version of the diabetes education/skills training materials every two weeks on the same schedule as the DM-CCT telephone sessions.
  Arms: Unconditional Cash Transfer-UCTs Intervention

SUMMARY:
This study will test the preliminary efficacy of diabetes-tailored CCT (DM-CCT), which will be conditional on participating in biweekly (every two weeks), nurse-led, virtual diabetes education/skills training and stress/coping intervention compared to UCT (with no requirement for participation) on clinical outcomes, self-care behaviors, and psychological health in 100 inner city AAs with poorly controlled T2DM using an RCT design. The aims of the proposed study include:

AIM 1: Test the preliminary efficacy of the DM-CCT intervention on glycemic control and quality of life for inner-city AAs with T2DM.

AIM 2: Test the preliminary efficacy of the DM-CCT intervention on self-care behaviors and psychological health for inner-city AAs with T2DM.

AIM 3: Estimate the cost of delivery of the DM-CCT and UCT interventions in preparation for future cost effectiveness analysis.

DETAILED DESCRIPTION:
The overarching aim of this proposal is to test the preliminary efficacy of diabetes-tailored CCT (DM-CCT conditional on participating in biweekly, nurse-led, virtual diabetes education/skills training and stress/coping intervention) compared to UCT (with no requirement for participation) on clinical outcomes, self-care behaviors, and psychological health in inner city African Americans with poorly controlled T2DM. One hundred (100) individuals will be randomized to either the DM-CCT intervention or the UCT intervention and followed for 6-months, with study visits at baseline, 3-months, and 6-months. The primary outcomes will be glycemic control (HbA1c) and quality of life (SF-12) at 6-months post randomization. The secondary outcomes will be self-care behaviors (diet, exercise, medication adherence) and psychological health (stress, coping) measured at 6-months post randomization. In preparation for future cost effectiveness studies, the final aim will estimate the cost of delivery of the DM-CCT and UCT interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Self-report as African American
* Clinical diagnosis of T2DM and HbA1c ≥8% at the screening visit
* Residence in inner city zip codes
* Income greater or equal to133% of federal poverty level or Medicaid eligible
* Able to communicate in English.

Exclusion Criteria:

* Mental confusion on interview suggesting significant dementia
* Alcohol or drug abuse/dependency
* Active psychosis or acute mental disorder
* Participation in other diabetes clinical trials
* Life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Glycemic control (HbA1c) | Change from baseline HbA1c at 6 months post intervention follow-ups
  Blood specimens (10cc of blood) will be obtained by trained phlebotomists or nurse for HbA1c.
Quality of Life as measured by SF-12 | Change from baseline quality of life measure at 6 months post intervention follow-ups
  The SF-12 (Ware 1996) is a valid and reliable instrument to measure functional status and reproduces 90% of the variance in PCS-36 and MCS-36 scores.

SECONDARY OUTCOMES:
Self-Care | Change from baseline self-care at 6 months post intervention follow-ups
  Behavioral skills will be assessed with the Summary of Diabetes Self-Care Activities (SDSCA) scale (Toobert 2000), a brief, validated questionnaire of diabetes self-care.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Campbell, PhD, Principal Investigator — State University at Buffalo
Locations (1):
- State University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers. Data may be available upon request in aggregate summary form.